CLINICAL TRIAL: NCT05302050
Title: A Cognitive Behavioral Digital Therapeutic InterventiON for Glycemic Control in Type 2 Diabetes Mellitus
Acronym: ACTION-DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Better Therapeutics (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM2-07-MGB
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study population consists of approximately 500 total participants, ages 18 - 75 years old, inclusive, who have type 2 diabetes. They will be randomized to the treatment or control group at a 3:1 ratio
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention BT-001 + Standard of Care (Active Comparator): Patients in this arm will receive the BT-001 treatment for up to 18 months.
  Interventions: Device: BT-001
- Standard of Care (Other): Patients will have access to a control mobile application for 6 months and then will have the option to use the treatment for the remainder of the 18 month study
  Interventions: Device: Control Mobile Application

INTERVENTIONS:
Device: BT-001 — BT-001is a software application that delivers treatment to participants with type 2 diabetes, using behavioral therapy. BT-001 is accessed via the participants' smartphone.
  The behavioral intervention process involves:
  Identifying maladaptive thoughts based on misinformed core beliefs that lead to disease-promoting behaviors; replacing maladaptive core beliefs with adaptive ways of thinking; and providing collaborative construction of behavioral exercises to test core beliefs.
  Each week, BT-001 asks participants to complete a new lesson, along with one skill exercise. The lessons are expected to take between 10-20 minutes to complete. In addition to completing a lesson and skill, participants will be directed to report plant-based meals consumed and minutes of exercise completed and to measure their blood sugar daily.
  Arms: Intervention BT-001 + Standard of Care
Device: Control Mobile Application — The app asks patients brief questions about their health but does not include any behavioral therapy.
  Arms: Standard of Care

SUMMARY:
Randomized, controlled, pragmatic trial with open-label extension evaluating BT-001, an investigational digital therapeutic intended to help patients with type 2 diabetes improve their glycemic control.

DETAILED DESCRIPTION:
The study intervention, BT-001 (the App), will be dispensed at enrollment to the Immediate Intervention App Use arm of the trial. Patients randomized to the Delayed Intervention App Use arm will be provided a "control App" with diabetes control, and then the BT-001 App after 180 days. Each participant is assigned to one 90-day treatment cycle of BT-001. Over the 12-month intervention period, study participants will be able to opt into up to 3 additional treatment cycles of BT-001. Study schema is included at the end of this section

ELIGIBILITY:
Inclusion Criteria:

* Current (within 3 months prior to enrollment) HbA1c >=7.01%
* Possession of and ability to use Android or iPhone mobile phone
* Speaks and reads in English
* Willing to measure frequent fasting finger glucose measurements as part of the App utilization

Exclusion Criteria:

* Current use of insulin other than a long-acting insulin analogue or human NPH insulin
* HbA1c >=11%
* Cognitive impairment or degenerative neuropsychiatric condition (e.g. Alzheimer's, dementia, mixed dementia, other significant memory loss, schizophrenia), or any other condition that in the Investigator's opinion may prevent patient from completing study activities
* Any terminal medical condition with life expectancy of < 1 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline and Day 180
  Change in HbA1c from baseline (enrollment) to 6 months after enrollment between groups.

SECONDARY OUTCOMES:
Change in HbA1c | Baseline and day 180, 365
  Change in HbA1c from baseline (enrollment) and from 6 months, to 12 months after enrollment between groups
Significant change in HbA1c | Baseline and Day 365
  Proportion of patients with a ≥ 0.4% decrease in HbA1c at 12 months within each study group

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham Hospital and Clinics, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared